CLINICAL TRIAL: NCT06609408
Title: The Effect of Nature and Game Based Activities on Happiness, Spiritual Well-Being, Frailty and Cognitive Status of Older People in Nursing Home
Brief Title: The Effect of Nature and Game Based Activities on Older People
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Murselcan Kabakcı, Specialist Nurse (PhD.), Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMU-2024-744
Record Dates: First submitted 2024-09-22; First posted 2024-09-24 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-09

CONDITIONS: Nature, Human; Older People; Nursing Home; Happiness; Spiritual Well-being; Frailty; Cognitive Ability, General
Keywords: Nature; Older People; Nursing Home; Happiness; Spiritual Well-Being; Frailty; Cognition
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Single blind randomised controlled mixed method trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Nature and game based activities will be applied to the participants in the experimental group once a week for 60 minutes for 8 weeks in this study.
  Interventions: Other: Nature and Game Based Activities
- Control Group (No Intervention): Individuals in the control group will not participate in the intervention. Individuals in control group will continue their routine activities in nursing home.

INTERVENTIONS:
Other: Nature and Game Based Activities — Individuals in experimental group will participate nature and game activities such as terrarium making, planting flowers, making puzzles in intervention.
  Arms: Experimental Group

SUMMARY:
The purpose of this study is determine the effect of nature and game based activities on happiness, spiritual well-being, frailty and cognitive status of older people in nursing home.

Hypotheses of the Research H0: Nature and game-based activities don't affect the happiness, spiritual well-being, cognitive function and frailty of older people in nursing home.

H1a: Happiness levels of older people in nursing home will be an increase after nature and game-based activities.

H1b: Spiritual well-being levels of older people in nursing home will be an increase after nature and game-based activities.

H1c: Cognitive function levels of older people in nursing home will be an increase after nature and game-based activities.

H1d: Frailty status of older people in nursing home will be a decrease after nature and game-based activities.

DETAILED DESCRIPTION:
The number and proportion of older people is increasing in the world and in Turkey. The number of older people is attracting more attention with the increase in older people health and rates. Ageing leads to an increase in chronic diseases and a decrease in physical functions, activities of daily living, independence, quality of life and general well-being. Older people transition from their living environment to institutions that provide long-term care such as nursing homes or retirement homes due to problems due to aging. The levels of happiness, spiritual well-being and cognitive function may decrease and the level of frailty may increase in older people staying in nursing homes. Various intervention methods are developed due to the increase in health care needs due to health problems occurring in older people in nursing homes. Nature and game based activities are non-pharmacological and low-risk intervention method that has the potential to increase physical, cognitive and psychological health levels and includes many activities. Gardening activities, which are an effective, individual oriented and nature based intervention method that focuses on improving the physical, cognitive, spiritual and emotional health aspects of older people in nursing homes. Gardening activity is supporting active and healthy ageing, provide a difference and innovation to the health services provided to older people receiving long term care. Gardening activity is an effective leisure activity and one of the easiest ways to provide easy access to green spaces. Older people who participate in gardening activities experience simple activities such as touching plants, smelling plants, tasting edible ones and many complex activities such as collecting seeds, sowing, planting, growing plants, cooking with harvested plants. Older people are positively influenced by emotional stimuli such as colours, smells, tastes, sights, sounds and grow products that can be very valuable for them in gardening activities. Experiences in nature is an opportunity to create spiritual meaning for the older people and contribute to the increase in the spiritual well-being levels of the older people. Gardening include different activities according to the functional ability levels of the participants such as manual dexterity and physical strength. Accordingly, gardening activities have the potential to improve the vulnerability of older people staying in nursing homes. Indoor gardening board game which is nature and game based activity are organised for older people who are limited in their daily life activities but can use their physical and cognitive functions. Individual characteristics, environment and weather conditions can affect the applicability of activities in open areas. Therefore, board games are independent of weather conditions and highly suitable activity to prevent cognitive impairments. Older people can easily access plant materials and actively interact with each other during board games. Thus memory, cognitive ability, motivation, speaking skills and social aspects are positively affected. In this context, nature and game based activities which are an effective and individual oriented intervention method contribute to the improvement of physical, cognitive, spiritual, emotional health aspects and support active and healthy ageing of older people in nursing homes. In addition, these activities provide diversity and innovation in health services provided to individuals receiving long-term care.

ELIGIBILITY:
Inclusion Criteria:

* Older people who have been in a nursing home for at least 6 months,
* Older people aged 65 years and over,
* Older people with a Mini Mental State score of 24 and above,
* Older people who are open to communication and co-operation will be included in the study.

Exclusion Criteria:

* Older people with physical problems that may prevent them from participating in nature and game based activities (such as stroke, Parkinson's),
* Older people with visual and hearing loss that may pose an obstacle to nature and game based activities,
* Older people with mental problems (such as dementia) that would prevent participation in nature and game based activities were excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Subjective Happiness Scale | This scale will be applied before and after the 8-week experiment.
  Subjective Happiness Scale was developed by Lyubomirsky and Lepper (1999) and adapted to Turkish by Akın and Satıcı (2011), and its validity and reliability were performed. This scale consists of 4 items in total and has a 7-point Likert type. The 4th item of the scale is reverse coded, and a total score is obtained by adding the scores of the items. A minimum of 4 and a maximum of 28 points are obtained from the scale. A high score from the scale indicates high perceived general subjective happiness, while a low score from the scale indicates low perceived subjective happiness. Cronbach Alpha coefficient of the scale is 0.86 and test-retest reliability coefficient is 0.73.
Standardized Mini Mental State Examination | This scale will be applied before and after the 8 weeks experiment.
  Standardized Mini Mental State Examination was developed by Folstein et al. (1975) to be used in dementia screening and adapted into Turkish by Güngen et al. (2002) to assess cognitive status. This scale is examined under five main headings and evaluated as recording memory (3 points), orientation (10 points), recall (3 points), attention and calculation (5 points) and language (9 points). There are two separate forms of the Mini Mental State for educated and uneducated individuals. The scale is evaluated out of 30 points; 24-30 is considered as normal, below 24 as cognitive impairment, 18-23 as mild dementia, 12-17 as moderate dementia and below 12 as severe dementia.
Tilburg Frailty Indicator | This scale will be applied before and after the 8-week experiment.
  Tilburg Frailty Indicator was developed by Gobbens et al. (2010) and adapted into Turkish and its validity and reliability was conducted by Arslan et al. (2018). Tilburg Frailty Scale consists of two parts. Part A includes 10 questions about diseases and sociodemographic factors that determine frailty; Part B consists of three factors that are components of frailty, including a total of 15 questions. The score range varies between 0-15; 5 or more a high score point is considered as frailty in Tilburg Frailty Indicator.
Spiritual Well-Being Scale | This scale will be applied before and after the 8-week experiment.
  Spiritual Well-Being Scale was developed by Ekşi and Kardaş (2017) for adults in order to determine the process of understanding and living their lives in personal, social, environmental and trascendental aspects in line with human values and ultimate meanings. The scale consists of 29 items and has a five-point Likert type. Seven questions in the scale (3, 7, 11, 15, 19, 23 and 26) are calculated inversely. The score that can be obtained from the scale is between 29-145. The higher the score obtained from the scale, the higher the level of spiritual well-being. Cronbach Alpha coefficient of the scale was found to be 0.886.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Aydın Avci, Prof. Dr., Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No